CLINICAL TRIAL: NCT02073357
Title: The BALANCED Anaesthesia Study A Prospective, Randomised Clinical Trial of Two Levels of Anaesthetic Depth on Patient Outcome After Major Surgery
Brief Title: The BALANCED Anaesthesia Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-1195
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Effect of General Anesthetic Dose on Recovery From Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Light general anaesthesia (BIS = 50) (Experimental): Light general anaesthesia
  Interventions: Procedure: Light general anaesthesia (BIS = 50)
- deep general anaesthesia (BIS = 35) (Experimental): deep general anaesthesia
  Interventions: Procedure: deep general anaesthesia (BIS = 35)

INTERVENTIONS:
Procedure: Light general anaesthesia (BIS = 50)
  Arms: Light general anaesthesia (BIS = 50)
Procedure: deep general anaesthesia (BIS = 35)
  Arms: deep general anaesthesia (BIS = 35)

SUMMARY:
General anaesthesia is a reversible drug-induced coma. Too little can result in patients being partially conscious during surgery; too much can slow recovery after surgery. There is a range of drug doses that can be used and some anesthesiologists use more than others. There is no convincing evidence that any particular dose within the usual range is better. Consequently, there are no guidelines on the best depth of anaesthesia. This study will determine whether general anesthetic concentrations at the low end of the usual range are better than those at the high end.

Participants will randomly be assigned to lighter or deeper general anesthesia. The first day after surgery, two short questionnaires about recovery and memories of the surgery will be completed. During the rest of the participant's hospital stay, a survey about how one feels will be completed.

There will be two telephone contacts after discharge from the hospital. One month after surgery three questionnaires will be completed about performing daily tasks, how you feel and memories of the surgery. Then one year after surgery pain will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years
* ASA physical status 3 or 4
* surgery expected to last ≥2 hours
* post-operative hospital stay expected to be ≥2 nights
* general anaesthesia with or without major regional block
* able to monitor BIS throughout anaesthesia

Exclusion Criteria:

* Unable to monitor BIS (e.g. cranial or intracranial surgery)
* unable to consent
* surgery with 'wake-up' test
* propofol infusion for part or all of maintenance of anaesthesia ('total intravenous anaesthesia')
* previous enrolment in Balanced study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
One-year all-cause mortality | One year

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sessler, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States